CLINICAL TRIAL: NCT00517751
Title: Treatment of Lumbar Spinal Stenosis With X-STOP® PEEK Spacer in Moderately Symptomatic Patients
Brief Title: Condition of Approval Study
Acronym: COAST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to Medtronic's voluntary withdrawal of PMA P040001 for X-STOP systems; post-approval study costs outweighed business benefits for marketing X-STOP in US.
Sponsor: Medtronic Spine LLC (Industry)
Responsible Party: Sponsor
Organization: Medtronic Spinal and Biologics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSS-006-COA
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2016-01

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar Spinal Stenosis; X-STOP Spacer; Interspinous process decompression; Neurogenic Intermittent Claudication
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- X-STOP PEEK (Experimental): In this arm, patients will undergo X-STOP PEEK surgery.
  Interventions: Device: X-STOP PEEK

INTERVENTIONS:
Device: X-STOP PEEK — Placement of X-STOP PEEK in up to two levels in the lumbar spine for patients diagnosed with moderately symptomatic lumbar spinal stenosis in accordance with current labeling instructions for use.

SUMMARY:
This prospective, multicenter longitudinal five-year study of X-STOP PEEK usage in LSS patients is designed to supplement pre-market safety and effectiveness data with information on longer-term device performance in a population of patients with moderately impaired physical function at preoperative baseline (i.e., an "indicated" population) who elect to undergo X STOP PEEK surgery.

DETAILED DESCRIPTION:
This prospective, multicenter longitudinal five-year study of X-STOP PEEK implant usage in LSS patients is designed to supplement pre-market safety and effectiveness data with information on longer-term device performance in a population of patients with moderately impaired physical function at preoperative baseline (i.e., an "indicated" population) who elect to undergo X-STOP PEEK surgery. This post-approval study will enroll 240 patients at up to 8 clinical sites where all participating spine surgeons have completed a company-sponsored physician training program. The clinical sites recruited to participate in this study comprise a geographically diverse mix of academic, referral, and/or community based sites.

Safety and effectiveness data will be assessed at baseline and annually through five (5) years postoperatively. Office visits will be scheduled preoperatively, and at 6 weeks, 1, 2, 3, 4, and 5 years postoperatively. Clinical/neurological and radiographic examination will be performed during each office visit. A baseline patient history (including medication usage) will be taken, and concomitant medications will be recorded at each postoperative follow-up visit. In addition, patients will be asked to complete the following questionnaires prior to consultation with their physicians or their staff: Zurich Claudication Questionnaire (ZCQ), Oswestry Disability Index (ODI), Numeric Rating Scale (NRS), and SF-36 Health Survey. At the 2-, 3-, 4- and 5-year office visit, patients will also be asked two questions assessing the value of surgery and the overall improvement in the quality of life postoperatively.

The primary study endpoint in this study is treatment success. Secondary endpoints will include scores from the SF-36, ODI, and NRS, as well as incidence rates of adverse events, device failures, and secondary surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. has a baseline score >2.0 in the Physical Function (PF) domain of the Zurich Claudication Questionnaire
2. is 50 years old or older
3. has leg/buttock/groin pain with or without back pain NOTE: Leg/buttock/groin pain must be completely relieved when flexed such as when sitting in a chair. If back pain is also present, it must be partially relieved when flexed.
4. can sit for 50 minutes without pain
5. can walk 50 feet or more
6. has a confirmed diagnosis of neurogenic intermittent claudication secondary to lumbar spinal stenosis, with X-Ray, MRI and/or CT evidence of thickened ligamentum flavum, narrowed lateral recess and/or central canal narrowing
7. has completed at least six months of conservative care therapy which may include but is not limited to physical therapy, bracing, systemic or injected medications
8. has signed a patient informed consent document
9. is physically and mentally willing and able or has a caregiver who can comply with the postoperative and routinely scheduled clinical and radiographic evaluations
10. lives in the immediate area and has no plans to relocate to another geographic area before completion of the study or lives outside the immediate area and will comply with the scheduled postoperative visits with a prearranged and designated physician

Exclusion Criteria:

1. has a baseline score less than or equal to 2.0 in the Physical Function (PF) domain of the Zurich Claudication Questionnaire
2. cannot sit for 50 minutes
3. cannot walk more than 50 feet
4. has unremitting pain in any spinal position
5. has axial back pain only without leg/buttock/groin pain
6. has a fixed motor deficit
7. has cauda equina syndrome defined as neural compression causing neurogenic bowel (rectal incontinence) or bladder (bladder retention or incontinence) dysfunction
8. has severe symptomatic lumbar spinal stenosis at more than two levels
9. has significant instability of the lumbar spine, e.g., isthmic spondylolisthesis or degenerative spondylolisthesis greater than grade 1 (on a scale of 1 to 4)
10. has an ankylosed segment at the affected level(s);
11. has significant scoliosis (Cobb angle is greater than 25 degrees)
12. has an acute fracture of the spinous process or pars interarticularis
13. has sustained pathologic fractures of the vertebrae or multiple fractures of the vertebrae and /or hips
14. has severe osteoporosis of the spine or hip, defined as bone mineral density (BMD) in the spine or hip more than 2.5 SD below the mean of adult normals in the presence of one or more fragility fractures
15. has Paget's disease at the involved segment(s) or metastasis to the vertebrae
16. has had any surgery of the lumbar spine
17. has significant peripheral neuropathy demonstrated by nerve conduction velocity tests
18. has acute denervation secondary to radiculopathy, as shown by EMG
19. has significant peripheral vascular disease characterized by diminished dorsalis pedus or tibial pulses
20. has extreme obesity as defined by a Body Mass Index (BMI) greater than 40 kg/m2
21. has an active systemic infection or infection localized to the site of implantation
22. has an active systemic disease such as AIDS, HIV, hepatitis, etc.
23. has a medical condition that may interfere with postoperative management and follow-up, or may result in patient death prior to study completion (e.g., Alzheimer's disease, unstable cardiac disease, active malignancy)
24. has a recent history of narcotic abuse (i.e., within last 3 years)
25. has a known allergy to titanium,titanium alloy, or polyetheretherketone
26. is immunologically suppressed, or has received or is receiving steroids at any dose daily for more than one month within the last 12 months
27. is currently involved in a study of another investigational product that may affect the outcome of this study
28. is pregnant or planning to become pregnant during the study period
29. cannot undergo MRI or tolerate closed MRI scanning.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2007-08; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Malcolm, MD, Principal Investigator — Pinnacle Orthopedics
Locations (23):
- United States (23):
  - The Kirklin Clinic - UAB Medical, Birmingham, Alabama
  - Tucson Orthopaedic Institute-East Office, Tucson, Arizona
  - Tucson Orthopaedic Institute-Northwest Office, Tucson, Arizona
  - Silicon Valley Spine Institute, Campbell, California
  - UC Davis Spine Center, Sacramento, California
  - UCLA Comprehensive Spine Center, Santa Monica, California
  - Colorado Neurosurgery Associates, P.C., Denver, Colorado
  - Panaorama Orthopedics and Spine Center, Golden, Colorado
  - Yale School of Medicine, Dept. of Orthopaedics, New Haven, Connecticut
  - George Washington University Hospital Medical Facility Associates, Washington D.C., District of Columbia
  - Pinnacle Orthopedics, Marietta, Georgia
  - Orthopaedic Center of Southern Illinois, Mount Vernon, Illinois
  - University of Kentucky, Dept of Neurosurgery, Lexington, Kentucky
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Drisko, Fee & Parkins, P.C., Kansas City, Missouri
  - UpState Orthopedics, East Syracuse, New York
  - Mayfield Clinic, Cincinnati, Ohio
  - The Center Orthopedic & Neurosurgical Care & Research, Bend, Oregon
  - NeuroSpine Institute, Eugene, Oregon
  - OrthopaediCare, Willow Grove, Pennsylvania
  - Texas Back Institute, Plano, Denton, Mansfield, Texas
  - Neurosurgical Associates of San Antonio, San Antonio, Texas
  - Scott & White Memorial Hospital & Scott, Sherwood & Brindley Foundation, Temple, Texas

REFERENCES:
- [Background] Zucherman JF, Hsu KY, Hartjen CA, Mehalic TF, Implicito DA, Martin MJ, Johnson DR 2nd, Skidmore GA, Vessa PP, Dwyer JW, Puccio ST, Cauthen JC, Ozuna RM. A multicenter, prospective, randomized trial evaluating the X STOP interspinous process decompression system for the treatment of neurogenic intermittent claudication: two-year follow-up results. Spine (Phila Pa 1976). 2005 Jun 15;30(12):1351-8. doi: 10.1097/01.brs.0000166618.42749.d1. PMID 15959362
- [Background] Hsu KY, Zucherman JF, Hartjen CA, Mehalic TF, Implicito DA, Martin MJ, Johnson DR 2nd, Skidmore GA, Vessa PP, Dwyer JW, Cauthen JC, Ozuna RM. Quality of life of lumbar stenosis-treated patients in whom the X STOP interspinous device was implanted. J Neurosurg Spine. 2006 Dec;5(6):500-7. doi: 10.3171/spi.2006.5.6.500. PMID 17176013
- [Background] Kondrashov DG, Hannibal M, Hsu KY, Zucherman JF. Interspinous process decompression with the X-STOP device for lumbar spinal stenosis: a 4-year follow-up study. J Spinal Disord Tech. 2006 Jul;19(5):323-7. doi: 10.1097/01.bsd.0000211294.67508.3b. PMID 16826002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to early study termination, the final analysis is consistent with the last annual report submission to the FDA and data reported on FDA's post-approval webpage reporting on 162 of 176 enrolled subjects.
Groups:
- X-STOP PEEK: In this arm, patients underwent X-STOP PEEK surgery.
Period: Overall Study
Arm/Group | X-STOP PEEK
Started | 162
Completed | 33
Not Completed | 129
Not completed — Death | 3
Not completed — Withdrawal by Subject | 37
Not completed — Lost to Follow-up | 4
Not completed — patient not over due | 6
Not completed — Patient not due for visit | 76
Not completed — Missing | 3

BASELINE CHARACTERISTICS:
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (8.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 87
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Black or African American | 4
  Hispanic or Latino | 4
  Native Hawaiian or other pacific islander | 1
  Caucasian | 152
  Other | 0
Height [Mean (Standard Deviation); unit: inches] | 67.2 (3.93)
Weight [Mean (Standard Deviation); unit: lbs] | 188.0 (37.40)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.3 (4.72)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success Rate at 24 Months
Description: Treatment success rate is reported as the percentage of participants who met all of the following criteria:
  1. Clinically significant improvement (by at least 0.5 points) in the Symptom Severity (SS) domain of the Zurich Claudication Questionnaire (ZCQ) compared to preoperative baseline
  2. Clinically significant improvement (by at least 0.5 points) in the Physical Function (PF) domain of the ZCQ compared to pre-operative baseline
  3. Patient satisfaction with treatment defined as a Patient Satisfaction (PS) score < 2.5
  4. No additional surgery for lumbar stenosis performed
  5. Maintenance of distraction
  6. No dislodgement of the implant
  7. No device-related complications
Time Frame: 24 months
Population: At 24 months, 94 subjects were evaluable for overall treatment success. Once subjects failed on additional surgery for lumbar stenosis or dislodgement of the implant or device-related complications, they failed at later visits no matter whether they had data or not.
Measure: Number; unit: percentage of participants
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 94
percentage of participants | 30.9

2. Secondary Outcome: Treatment Success Rate at 60 Months
Description: Treatment success rate is reported as the percentage of participants who met all of the following criteria:
  1. Clinically significant improvement (by at least 0.5 points) in the Symptom Severity (SS) domain of the ZCQ compared to preoperative baseline
  2. Clinically significant improvement (by at least 0.5 points) in the Physical Function (PF) domain of the ZCQ compared to pre-operative baseline
  3. Patient satisfaction with treatment defined as a Patient Satisfaction (PS) score < 2.5
  4. No additional surgery for lumbar stenosis performed
  5. Maintenance of distraction
  6. No dislodgement of the implant
  7. No device-related complications
Time Frame: 60 months
Population: At 60 months, 62 subjects were evaluable for overall treatment success. Once subjects failed on additional surgery for lumbar stenosis or dislodgement of the implant or device-related complications, they failed at later visits no matter whether they had data or not.
Measure: Number; unit: percentage of participants
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 62
percentage of participants | 24.2

3. Secondary Outcome: Symptom Severity (SS) Scores Measured by Zurich Claudication Questionnaire (ZCQ)
Description: ZCQ is a validated outcomes instrument specific to lumbar spinal stenosis, and captures data in 3 distinct domains: SS, PF, and post-treatment PS. SS Score is based on seven questions (overall pain, pain frequency, pain in the back, pain in the leg, numbness, weakness, and balanced disturbance) in ZCQ. The first 6 questions are scored 1 to 5. Balance disturbance is scored in a 1-3-5 scale. The SS score is the mean of all answered items in the questionnaire, ranging from 1 to 5. A lower score represents a better outcome/condition. If more than two items were missing, the SS score was considered as missing.
Time Frame: Baseline, 6 weeks, 12 months, 24 months, 36 months, 48 months, and 60 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
units on a scale
  SS score baseline (n=161) | 3.29 (0.58)
  SS score at 6 weeks (n=151) | 2.10 (0.70)
  SS score at 12 months (n=103) | 2.26 (0.77)
  SS score at 24 months (n=88) | 2.38 (0.85)
  SS score at 36 months (n=71) | 2.25 (0.78)
  SS score at 48 months (n=59) | 2.32 (0.81)
  SS score at 60 months (n=46) | 2.38 (0.89)

4. Secondary Outcome: Success Rate in Symptom Severity (SS) Domain of Zurich Claudication Questionnaire (ZCQ)
Description: Success rate in SS domain of ZCQ is reported as percentage of participants who had success in SS domain of the ZCQ. The SS success was defined as clinically significant improvement by at least 0.5 point in SS score compared to preoperative baseline.
Time Frame: 6 weeks, 12months, 24 months, 36 months, 48 months, and 60 months
Measure: Number; unit: percentage of participants
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
percentage of participants
  SS success at 6 weeks (n=150) | 78.0
  SS success at 12 months (n=102) | 71.6
  SS success at 24 months (n=87) | 62.1
  SS success at 36 months (n=70) | 64.3
  SS success at 48 months (n=59) | 61.0
  SS success at 60 months (n=46) | 56.5

5. Other Pre Specified Outcome: Percent of Subjects With Pfirrmann Grades Increased From Baseline at Any Index Level at 24 Months
Description: The Pfirrmann Grading System is descriptive and grades the status on an intervertebral disc as visualized with MRI using a 5-point system (grade I, II, III, IV or V). Grade I: disc is homogeneous with bright hyper-intense white signal intensity and normal disc height. Grade V: disc is inhomogeneous with hypo-intense black signal intensity and there is no more distinction between the nucleus and annulus, the disc space is collapsed. The percent of subjects with Pfirrmann grades increased from baseline at 24 months is reported.
Time Frame: 24 months
Population: At 24 months, 53 subjects were evaluable for Pfirrmann Grade assessment.
Measure: Number; unit: percentage of participants
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 53
percentage of participants | 9.4

6. Other Pre Specified Outcome: Percent of Subjects With Pfirrmann Grades Increased From Baseline at Any Index Level at 60 Months
Description: The Pfirrmann Grading System is descriptive and grades the status on an intervertebral disc as visualized with MRI using a 5-point system (grade I, II, III, IV or V). Grade I: disc is homogeneous with bright hyper-intense white signal intensity and normal disc height. Grade V: disc is inhomogeneous with hypo-intense black signal intensity and there is no more distinction between the nucleus and annulus, the disc space is collapsed. The percent of subjects with Pfirrmann grades increased from baseline at 60 months is reported.
Time Frame: 60 months
Population: At 60 months, 16 subjects were evaluable for Pfirrmann Grade assessment.
Measure: Number; unit: percentage of participants
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 16
percentage of participants | 0.0

7. Other Pre Specified Outcome: Percent of Subjects With Pfirrmann Grades Increased at Adjacent Levels at 24 Months
Description: The percent of subjects with Pfirrmann grades increased from baseline at adjacent levels at 24 months is reported.
Time Frame: 24 months
Population: At 24 months, 53 subjects were evaluable for Pfirrmann Grade assessment.
Measure: Number; unit: percentage of participants
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 53
percentage of participants | 9.4

8. Secondary Outcome: Physical Function (PF) Scores Measured by Zurich Claudication Questionnaire (ZCQ)
Description: PF score is the mean score of five physical function questions of ZCQ, ranging from 1 to 4. A lower score represents a better outcome/condition. If more than one item were missing, the PF score was considered as missing.
Time Frame: Baseline, 6 weeks, 12 months, 24 months, 36 months, 48 months, and 60 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
units on a scale
  PF score at baseline (n=162) | 2.67 (0.36)
  PF score at 6 weeks (n=150) | 1.79 (0.60)
  PF score at 12 months (n=103) | 1.71 (0.62)
  PF score at 24 months (n=87) | 1.89 (0.69)
  PF score at 36 months (n=71) | 1.93 (0.76)
  PF score at 48 months (n=59) | 1.87 (0.67)
  PF score at 60 months (n=46) | 1.92 (0.79)

9. Secondary Outcome: Success Rate in Physical Function (PF) Domain of Zurich Claudication Questionnaire (ZCQ)
Description: Success rate in PF domain of ZCQ is reported as percentage of participants who had success in PF domain of ZCQ. The PF success was defined as clinically significant improvement by at least 0.5 points in PF score compared to preoperative baseline.
Time Frame: 6 weeks, 12months, 24 months, 36 months, 48 months, and 60 months
Measure: Number; unit: percentage of participants
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
percentage of participants
  PF success at 6 weeks (n=150) | 70.7
  PF success at 12 months (n=103) | 71.8
  PF success at 24 months (n=87) | 59.8
  PF success at 36 months (n=71) | 56.3
  PF success at 48 months (n=59) | 61.0
  PF success at 60 months (n=46) | 54.3

10. Secondary Outcome: Patient Satisfaction (PS) Scores Measured by Zurich Claudication Questionnaire (ZCQ) at Post Treatment
Description: PS score is the mean score of 6 questions of ZCQ, ranging from 1 to 4 if the number of responses exceeded four. A lower score represents a better outcome. Patients with PS score less than 2.5 at postoperative evaluation were considered positive, which implied that patients were satisfied with their treatment.
Time Frame: 6 weeks, 12 months, 24 months, 36 months, 48 months, and 60 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
units on a scale
  PS score at 6 weeks (n=150) | 1.75 (0.74)
  PS score at 12 months (n=103) | 1.78 (0.75)
  PS score at 24 months (n=88) | 1.90 (0.81)
  PS score at 36 months (n=70) | 1.84 (0.81)
  PS score at 48 months (n=59) | 1.89 (0.90)
  PS score at 60 months (n=46) | 1.91 (0.90)

11. Secondary Outcome: Success Rate in Patient Satisfaction (PS) Domain of Zurich Claudication Questionnaire (ZCQ) at Post Treatment
Description: Success rate in PS domain of ZCQ at post treatment is reported as the percentage of participants who had success in PS domain of ZCQ. The PS success was defined as PS score less than 2.5.
Time Frame: 6 weeks, 12months, 24 months, 36 months, 48 months, and 60 months
Measure: Number; unit: percentage of participants
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
percentage of participants
  PS success at 6 weeks (n=150) | 81.3
  PS success at 12 months (n=103) | 80.6
  PS success at 24 months (n=88) | 72.7
  PS success at 36 months (n=70) | 72.9
  PS success at 48 months (n=59) | 67.8
  PS success at 60 months (n=46) | 69.6

12. Secondary Outcome: Oswestry Disability Index (ODI) Score
Description: ODI Questionnaire was used to assess patient back function. The ODI score ranges from 0-100. The best score is 0 (no disability) and worst is 100 (maximum disability).
Time Frame: Baseline, 6 weeks, 12 months, 24 months, 36 months, 48 months, and 60 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
units on a scale
  ODI score at baseline (n=162) | 38.81 (14.11)
  ODI score at 6 weeks (n=151) | 22.98 (16.23)
  ODI score at 12 months (n=103) | 20.34 (16.27)
  ODI score at 24 months (n=88) | 23.99 (17.08)
  ODI score at 36 months (n=71) | 23.04 (17.23)
  ODI score at 48 months (n=59) | 25.27 (18.22)
  ODI score at 60 months (n=46) | 24.88 (18.53)

13. Secondary Outcome: General Health Status -- SF-36 PCS
Description: The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) was used to assess general health status. The SF-36 results were summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The score for PCS is between 0 and 100, with higher scores denoting better quality of life.
Time Frame: Baseline, 6 weeks, 12 months, 24 months, 36 months, 48 months, and 60 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
units on a scale
  SF-36 PCS at baseline (n=162) | 27.1 (6.8)
  SF-36 PCS at 6 week (n=150) | 36.3 (10.5)
  SF-36 PCS at 12 months (n=103) | 38.4 (12.2)
  SF-36 PCS at 24 months (n=88) | 35.2 (12.0)
  SF-36 PCS at 36 months (n=70) | 36.4 (12.5)
  SF-36 PCS at 48 months (n=58) | 35.7 (11.8)
  SF-36 PCS at 60 months (n=46) | 35.6 (12.6)

14. Secondary Outcome: General Health Status -- SF-36 MCS
Description: MCS score is between 0 and 100, with higher scores denoting better quality of life.
Time Frame: Baseline, 6 weeks, 12 months, 24 months, 36 months, 48 months, and 60 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
units on a scale
  SF-36 MCS at baseline (n=162) | 51.5 (10.8)
  SF-36 MCS at 6 weeks (n=150) | 54.6 (9.5)
  SF-36 MCS at 12 months (n=103) | 53.8 (10.1)
  SF-36 MCS at 24 months (n=88) | 53.4 (11.1)
  SF-36 MCS at 36 months (n=70) | 54.6 (10.8)
  SF-36 MCS at 48 months (n=58) | 54.1 (11.9)
  SF-36 MCS at 60 months (n=46) | 52.8 (12.5)

15. Other Pre Specified Outcome: Percent of Subjects With Pfirrmann Grades Increased at Adjacent Levels at 60 Months
Description: The percent of subjects with Pfirrmann grades increased from baseline at adjacent levels at 60 months is reported.
Time Frame: 60 months
Population: At 60 months, 16 subjects were evaluable for Pfirrmann Grade assessment.
Measure: Number; unit: percentage of participants
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 16
percentage of participants | 25.0

16. Secondary Outcome: Back Pain in Numerical Rating Scales (NRS)
Description: Back pain was measured using NRS. Patients rated their back pain on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be."
Time Frame: Baseline, 6 weeks, 12 months, 24 months, 36 months, 48 months, and 60 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
units on a scale
  Back pain at baseline (n=161) | 6.4 (2.4)
  Back pain at 6 weeks (n=150) | 3.2 (2.4)
  Back pain at 12 months (n=103) | 3.5 (2.8)
  Back pain at 24 months (n=88) | 4.0 (3.0)
  Back pain at 36 months (n=70) | 3.7 (2.9)
  Back pain at 48 months (n=59) | 3.7 (3.2)
  Back pain at 60 months (n=46) | 3.5 (3.0)

17. Secondary Outcome: Left Leg Pain in Numerical Rating Scales (NRS)
Description: Left leg pain was measured using NRS. Patients rated their leg pain on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be."
Time Frame: Baseline, 6 weeks, 12 months, 24 months, 36 months, 48 months, and 60 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
units on a scale
  Left leg pain at baseline (n=161) | 5.5 (3.0)
  Left leg pain at 6 weeks (n=150) | 1.9 (2.6)
  Left leg pain at 12 months (n=103) | 2.1 (2.8)
  Left leg pain at 24 months (n=87) | 2.7 (2.9)
  Left leg pain at 36 months (n=70) | 2.8 (3.0)
  Left leg pain at 48 months (n=59) | 2.5 (2.9)
  Left leg pain at 60 months (n=46) | 2.7 (3.1)

18. Secondary Outcome: Right Leg Pain in Numerical Rating Scales (NRS)
Description: Right leg pain was measured using NRS. Patients rated their leg pain on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be."
Time Frame: Baseline, 6 weeks, 12 months, 24 months, 36 months, 48 months, and 60 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
units on a scale
  Right leg pain at baseline (n=161) | 5.5 (3.0)
  Right leg pain at 6 weeks (n=150) | 2.0 (2.5)
  Right leg pain at 12 months (n=103) | 2.4 (2.7)
  Right leg pain at 24 months (n=88) | 2.9 (3.1)
  Right leg pain at 36 months (n=70) | 2.3 (2.7)
  Right leg pain at 48 months (n=59) | 2.7 (3.2)
  Right leg pain at 60 months (n=46) | 2.8 (3.2)

19. Other Pre Specified Outcome: Percent of Subjects Who Reported Implant-Related Adverse Events
Time Frame: Overall study period
Measure: Number; unit: percentage of participants
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
percentage of participants | 11.1

20. Other Pre Specified Outcome: Percent of Subjects Who Had Any Subsequent Lumbar Spine Surgery
Time Frame: Overall study period
Measure: Number; unit: percentage of participants
Arm/Group | X-STOP PEEK
Number analyzed (Participants) | 162
percentage of participants | 19.8

ADVERSE EVENTS:
Time Frame: Overall study period (up to 60 months)
Description: Due to early study termination, not all subjects were followed through 60 months.
Arm/Group | X-STOP PEEK
Serious Adverse Events (participants affected / at risk) | 65/162
Other Adverse Events (participants affected / at risk) | 118/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | X-STOP PEEK (N=162)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3)
Diastolic dysfunction (Cardiac disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Myocarditis (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Haematotympanum (Ear and labyrinth disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Cataract cortical (Eye disorders) | 1 (1)
Macular hole (Eye disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal fissure (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Death (General disorders) | 2 (2)
Device dislocation (General disorders) | 3 (3)
Device ineffective (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Medical device pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 2 (2)
Meningitis bacterial (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Post procedural infection (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 2 (3)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Cardiac stress test abnormal (Investigations) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Total fluid volume decreased (Metabolism and nutrition disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (4)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 (3)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 3 (3)
Cervical myelopathy (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Intracranial hypotension (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 2 (2)
Radiculopathy (Nervous system disorders) | 2 (2)
Sensory disturbance (Nervous system disorders) | 1 (1)
Spinal claudication (Nervous system disorders) | 9 (9)
Delusion (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Activities of daily living impaired (Social circumstances) | 2 (2)
Abdominal hernia repair (Surgical and medical procedures) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1)
External fixation of fracture (Surgical and medical procedures) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Joint dislocation reduction (Surgical and medical procedures) | 1 (1)
Leg amputation (Surgical and medical procedures) | 1 (1)
Medical device removal (Surgical and medical procedures) | 20 (22)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Iliac artery thrombosis (Vascular disorders) | 1 (2)
Vascular insufficiency (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | X-STOP PEEK (N=162)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2)
Diastolic dysfunction (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3)
Cataract nuclear (Eye disorders) | 1 (1)
Corneal bleeding (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Faecal incontinence (Gastrointestinal disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal infection (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Levator syndrome (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Adverse drug reaction (General disorders) | 4 (4)
Asthenia (General disorders) | 1 (1)
Axillary pain (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Complication of device insertion (General disorders) | 5 (5)
Device difficult to use (General disorders) | 1 (1)
Device dislocation (General disorders) | 3 (3)
Device material issue (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Gait disturbance (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 2 (3)
Pyrexia (General disorders) | 1 (1)
Xerosis (General disorders) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4)
Candidiasis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 5 (5)
Incision site infection (Infections and infestations) | 3 (3)
Influenza (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 2 (2)
Laryngitis viral (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (7)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Urinary tract infection (Infections and infestations) | 6 (11)
Wound infection staphylococcal (Infections and infestations) | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1)
Dural tear (Injury, poisoning and procedural complications) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 18 (23)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 2 (2)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Incision site oedema (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 8 (8)
Incision site pruritus (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2)
Operative haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (2)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 4 (4)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 8 (8)
Tendonitis (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 5 (6)
Blood glucose increased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 3 (3)
Blood triglycerides increased (Investigations) | 2 (2)
Body temperature increased (Investigations) | 1 (1)
Glysolated haemoglobin increased (Investigations) | 1 (1)
Pulse absent (Investigations) | 1 (1)
Spinal x-ray abnormal (Investigations) | 1 (1)
Weight decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (21)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 35 (49)
Bursitis (Musculoskeletal and connective tissue disorders) | 6 (6)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (2)
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 (5)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 (13)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (13)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 11 (11)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 (12)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (19)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (4)
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (4)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Amnesia (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 2 (3)
Cerebral atrophy (Nervous system disorders) | 1 (1)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (1)
Coordination abnormal (Nervous system disorders) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 6 (9)
Lethargy (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 2 (2)
Multiple sclerosis (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (4)
Poor quality sleep (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Radicular pain (Nervous system disorders) | 5 (5)
Senile dementia (Nervous system disorders) | 1 (1)
Spinal claudication (Nervous system disorders) | 8 (12)
Tarsal tunnel syndrome (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Flashback (Psychiatric disorders) | 1 (1)
Grief reaction (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Sleep disorder (Psychiatric disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (2)
Nocturia (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Strangury (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysponea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 4 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Corneal transplant (Surgical and medical procedures) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Peripheral coldness (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Study strengths include collection of 5-year data and radiographic examinations. Study weaknesses include single-arm design and early termination of the study without reaching the desired sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less